CLINICAL TRIAL: NCT06887088
Title: Phase II, Single Arm, Multicentre Clinical Trial to Evaluate the Activity of Encorafenib Plus Binimetinib Followed by Cemiplimab And Fianlimab in Patients With BRAF Mutated Melanoma and Symptomatic Brain Metastases
Brief Title: Encorafenib and biNimetinib Followed by CEmiplimab and FiAnLimab in Patients With BRAF Mutant melanOma and Symptomatic Brain Metastases
Acronym: ENCEFALO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); MFAR (Other); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-2301; 2024-513375-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Melanoma BRAF V600E/K Mutated; Melanoma and Brain Metastases
Keywords: Melanoma; Encorafenib; Binimetinib; Cemiplimab; Fianlimab; BRAF mutant
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: ENCEFALO is a multicentre, single arm phase II clinical trial in patients with melanoma BRAF-mutated and symptomatic brain metastases that follows Simon Two Stages Minimax design.
  The trial will enroll competitively up to 33 patients. The study will enroll the first 18 patients and monitor for progression at 6 months (24-weeks assessment). If there are 4 or less patients free of progression at the 6-months tumor assessment the accrual will be closed. Otherwise, a minimum of 15 additional patients will be accrued for a total of 33 evaluable patients. All patients will have a histologically confirmed diagnosis of unresectable metastatic BRAF-mutated melanoma, with one or more brain metastases with a diameter of 5 to 50 mm and symptomatology associated with the disease, defined as symptom related with intracranial hypertension or cognitive impairment. all patients will be ≥ 18 years and ECOG PS 0-2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Encorafenib+biNimetinib followed Cemiplimab+Fianlimab in BRAF mutated melanoma and brain metastses (Experimental): Patients with BRAF mutant melanoma and symptomatic brain metastases will treatment with encorafenib plus binimetinib followed by cemiplimab and fianlimab Induction treatment with oral encorafenib 450 mg once daily (QD) + binimetinib 45 mg twice daily (BID)(combination: EB) for approximately two months (i.e. 8 weeks) followed by cemiplimab 350 mg + fianlimab 1600 mg combination every 3 weeks (Q3W)(Combination: CF) administered to patients intravenously (IV) for up to two years. Treatment may be discontinued due to death, PD or non-acceptable toxicity. Encorafenib plus binimetinib should be discontinued at least 72 hours prior to the first dose of cemiplimab plus fianlimab. Rechallenge with encorafenib 450mg QD + binimetinib 45 mg BID will be mandatory for those patients that progress under CF, with the exception of patients with intracranial response or stabilization and only extracranial PD in which case CF could be continued at the physician criteria. In the case of continuing treat
  Interventions: Drug: Encorafenib + Binimetinib; Drug: cemiplimab+fianlimab

INTERVENTIONS:
Drug: Encorafenib + Binimetinib — Induction treatment with oral encorafenib 450 mg once daily (QD) + binimetinib 45 mg twice daily (BID)(combination: EB) for approximately two months (i.e. 8 weeks)
Drug: cemiplimab+fianlimab — cemiplimab 350 mg + fianlimab 1600 mg combination every 3 weeks (Q3W)(Combination: CF) administered to patients intravenously (IV) for up to two years.

SUMMARY:
Brain metastases in patients with advanced and metastatic melanoma are a frequent complication and a significant cause of morbidity and mortality in this patient population. As the incidence of brain metastases continues to increase in patients with metastatic melanoma, it is urgent that the investigators identify effective therapies.

ENCEFALO is a Phase II, single arm, multicentre clinical trial designed to evaluate the activity of encorafenib plus binimetinib followed by cemiplimab and fianlimab in patients with BRAF mutated melanoma and symptomatic brain metastases, following the simon design Two-stage minimax.

The objective main is to evaluate the 6 month intracranial progression-free survival (icPFS) proportion of Encorafenib plus Binimetinib followed by Cemiplimab plus Fianlimab in patients with BRAF-mutated melanoma and symptomatic brain metastases according RECIST criteria

The trial hypothesis is: For patients with BRAF-mutated melanoma and symptomatic brain metastases, an induction treatment with encorafenib and binimetinib (EB) for about two months (i.e. 8 weeks) followed by cemiplimab plus fianlimab (CF) would allow a 6 month icPFS rate of 40% in comparison to historical control of 20% based on CM204 symptomatic arm (Tawbi et al 2021).

DETAILED DESCRIPTION:
1. RATIONAL

   Melanoma with Brain Metastasis Background

   Brain metastases in patients with advanced and metastatic melanoma are a frequent complication and a significant cause of morbidity and mortality in this patient population. As the incidence of brain metastases continues to increase in patients with metastatic melanoma, it is urgent that the investigators identify effective therapies.

   Recent data have shown an incidence of brain metastases in ≤ 50% of patients with metastatic melanoma (Chukwueke U et al 2016). Because this is typically a late complication of systemic disease, melanoma-related brain metastases have been associated with significant neurologic morbidity and a poor median overall survival, with treatment, of approximately 9 months (Ramanujam S et al 2015). Factors that predict survival include age, performance status, and the number of brain metastases, which are summarized as the melanoma-specific graded prognostic assessment (Sperduto PW et al 2010).

   Systemic Therapy for Melanoma Patients with Brain Metastases

   Patients with BRAF-mutated melanoma and symptomatic brain metastases (SBM) have a high unmet medical need. On one hand, treatment with ipilimumab and nivolumab yields the best results in patients with asymptomatic disease, according to CM204 and ABC studies (Tawbi HA et al 2021)(Long GV et al 2021), but it has worse outcomes for patients with symptomatic disease, according to CM204 study (Tawbi HA et al 2021). On the other hand, targeted therapy with dabrafenib and trametinib yields a high response rate that is independent of the symptomatic status (Davies MA et al 2017) although the durability of these responses is usually short termed, in contrast with immunotherapy (Davies MA et al 2017).

   A phase I clinical trial has demonstrated a promising maintained activity with the combination of cemiplimab and fianlimab in patients with unresectable or metastatic melanoma who were all naïve to anti-PD-1 therapy for advanced disease (n=98). The ORR was 61%, the median progression-free survival (PFS) was 15 months (Hamid O et al 2023). The combination is currently being investigated in patients with melanoma at diverse stages (Baramidze A et al 2023)(Panella TJ et al 2023). Additionally, the relativity clinical trial has demonstrated an improvement of PFS with the combination of nivolumab and relatlimab in comparison to nivolumab (Tawbi HA et al 2022), although patients with brain metastases were underrepresented.

   In addition, a previous communication suggests that the treatment with immunotherapy is not as efficacious for patients with BRAF-mutated melanoma and brain metastases previously treated and progressed to targeted therapy (Lau PKH et al 2021).

   The sandwich approach (starting with targeted therapy based in encorafenib and binimetinib followed by dual immune checkpoint blockade without waiting to progression) has been demonstrated that sequencing targeted and immunotherapy is a feasible strategy in the SECOMBIT clinical trial (Ascierto PA et al 2021).

   Recetly, the Spanish Melanoma Group (GEM) has published the results of the EBRAIN/GEM1802 clinical trial, evaluates the treatment with encorafenib and binimetinib (EB) followed by radiotherapy in symptomatic and asymtomatic patients with BRAF mutated melanoma and brain metastases, showing and intracranial objective response of 70.8% and complete response of 10.4%. This clinical trial also explores if radiotherapy after achieving an objective response or stable disease in the brain could improve the intracranial progression free survival (icPFS). Median icPFS and OS were 8.5 and 15.9 months, respectively (8.3 months for icPFS and 13.9 months OS for patients receiving radiotherapy). In conclusion, encorafenib plus binimetinib showed promising clinical benefit in terms of icRR and tolerable safety profile. Sequential radiotherapy is feasible but it does not seem to prolong response (Marquez-Rodas I et al 2024).
2. HYPOTHESIS For patients with BRAF-mutated melanoma and symptomatic brain metastases, an induction treatment with encorafenib and binimetinib (EB) for about two months (i.e. 8 weeks) followed by cemiplimab plus fianlimab (CF) would allow a 6 month icPFS rate of 40% in comparison to historical control of 20% based on CM204 symptomatic arm (Margolin KA et al 2021).
3. STUDY TREATMENTS Induction treatment with oral encorafenib 450 mg once daily (QD) + binimetinib 45 mg twice daily (BID)(combination: EB) for approximately two months (i.e. 8 weeks) followed by cemiplimab 350 mg + fianlimab 1600 mg combination every 3 weeks (Q3W)(Combination: CF) administered to patients intravenously (IV) for up to two years. Treatment may be discontinued due to death, PD or non-acceptable toxicity. Encorafenib plus binimetinib should be discontinued at least 72 hours prior to the first dose of cemiplimab plus fianlimab. Rechallenge with encorafenib 450mg QD + binimetinib 45 mg BID will be mandatory for those patients that progress under CF, with the exception of patients with intracranial response or stabilization and only extracranial PD in which case CF could be continued at the physician criteria. In the case of continuing treatment with CF, tumor assessment should be repeated after 8 weeks to confirm the progression and the benefit of CF to the brain.
4. OBJECTIVES Primary Objectives To evaluate the 6 month intracranial progression-free survival (icPFS) proportion of Encorafenib plus Binimetinib followed by Cemiplimab plus Fianlimab in patients with BRAF-mutated melanoma and symptomatic brain metastases.

   Secondary Efficacy Objectives

   To assess the following efficacy endpoints:
   * 12 month icPFS rate
   * Intracraneal PFS (icPFS)
   * Extracraneal PFS (ecPFS)
   * Global PFS (PFS)
   * Overall survival (OS)
   * Intracranial objective response rate (icORR) at 2 and 6 months
   * Extracraneal ORR (ecORR) at 2 and 6 months
   * Basal Quality of Life (QoL), at 2 and 6 months
   * Basal systemic steroids decrease at 2 and 6 months
   * Modified Barthel index improvement at 2 and 6 months Secondary Safety Objectives To assess the following the safety profile of the combination through continuous assessment of Adverse events (AE) and Treatment-related AEs (TRAEs).

   Secondary Exploratory Objectives To evaluate the correlation between biomarkers and the clinical outcomes of treatment with encorafenib plus binimetinib followed by cemiplimab plus fianlimab in patients with BRAF-mutated melanoma and symptomatic brain metastases.
5. ENDPOINTS The primary endpoint for ENCEFALO is the 6 month intracranial progression-free survival (icPFS), defined as the proportion of patients alive and free of icPFS according to modified RECIST criteria at 6 month evaluation (week 24 +/- 3 weeks) after the start of study treatment. The icPFS will be assessed locally by investigators.

   Secondary Efficacy Endpoints
   * 12-months icPFS: Percentage of patients free of icPFS according to modified RECIST criteria at 12 month evaluation (week 48 +/- 3 weeks).
   * icPFS locally assessed according to modified RECIST criteria, median and global curve estimated by kaplan meier method
   * ecPFS locally assessed according to modified RECIST criteria, median and global curve estimated by kaplan meier method
   * PFS locally assessed according to modified RECIST criteria, median and global curve estimated by kaplan meier method
   * OS locally assessed, median and global curve estimated by kaplan meier method
   * Change in patient reported outcomes in Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3.
   * Changes in Barthel score from baseline.
   * Change in systemic steroids usage from baseline. Secondary Safety Endpoints

   Type, incidence, frequency, severity and relation to the treatment of reported adverse events, physical examinations and laboratory tests:
   * Frequency and severity of adverse events assessed by NCI CTCAE v5.0.
   * Frequency of treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0.
   * Frequency of AEs leading to treatment discontinuation. Secondary Exploratory Endpoints
   * Expression of circulating tumor DNA (ctDNA) in blood samples at several time points throughout the study treatment.
   * Presence of peripheral blood mononuclear cells (PMDCs) in blood samples at several time points throughout the study treatment.
6. STUDY DESIGN

   The trial will enroll competitively up to 33 patients. The study will enroll the first 18 patients and monitor for progression at 6 months (24-weeks assessment). If there are 4 or less patients free of progression at the 6-months tumor assessment the accrual will be closed. Otherwise, a minimum of 15 additional patients will be accrued for a total of 33 evaluable patients. All patients will have a histologically confirmed diagnosis of unresectable metastatic BRAF-mutated melanoma, with one or more brain metastases with a diameter of 5 to 50 mm and symptomatology associated with the disease, defined as symptom related with intracranial hypertension or cognitive impairment. all patients will be ≥ 18 years and ECOG PS 0-2 (See Section 8 for further detail on eligibility).

   The design includes a screening phase in which patient eligibility is addressed, a treatment phase, and a follow-up phase.

   Study treatment will begin as soon as possible after signing the informed consent and inclusion will be completed as is indicated in protocol.

   All enrolled patients will receive an induction treatment with oral encorafenib 450 mg once daily (QD) + binimetinib 45 mg twice daily (BID)(combination: EB) for approximately two months (i.e. 8 weeks) followed by cemiplimab 350 mg + fianlimab 1600 mg combination every 3 weeks (Q3W)(Combination: CF) administered to patients intravenously (IV) for up to 2 years. Treatment may be discontinued due to death, PD or non-acceptable toxicity

   . Rechallenge with encorafenib 450mg QD + binimetinib 45 mg BID will be mandatory for those patients that progress under CF, with the exception of patients with intracranial response or stabilization and only extracranial PD in which case CF could be continued at the physician criteria. In the case of continuing treatment with CF, tumor assessment should be repeated after 8 weeks, and no longer, to confirm the progression and the brain benefit.

   The primary endpoint is efficacy determined by the 6-month icPFS proportion. All patients will undergo periodic mandatory tumor assessments by CT or MRI scan every 8 weeks ± 7 days for the first year from the start of study treatment and recommended every 12 weeks ± 7 days afterwards until progression or patient withdrawal. Further CT/MRI scans could be performed upon suspicion of disease progression according to standard clinical practice and physician criteria. Safety will be assessed at every visit through continuous monitoring of signs and symptoms and periodic laboratory analysis.
7. SAMPLE SIZE Using Simon's two-stage Minimax design (Simon R 1989), assuming the null hypothesis as the rate of patients not progressing in the brain at 6 months (defined as a success) is about 20% (Tawbi et al. 2021), will be tested against a one-sided alternative (40%). In the first stage Simon's two-stage minimax design, 18 patients will be accrued. If there are ≤4 successes (defined as patients not progressing at 6 months) in these 18 patients, the study will be stopped. Otherwise, a minimum of 15 additional patients will be accrued for a total of 33 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all the following criteria:

* Written informed consent approved by the Independent Ethics Committee (IEC), prior to the performance of any trial activities.
* Histologically confirmed diagnosis of unresectable metastatic BRAF-mutated melanoma (stage IV, AJCC v9), with one or more brain metastases with a diameter of 5 to 50 mm, measured by contrast enhanced MRI.
* Patients with brain metastasis that debut as symptomatic, regardless of corticosteroid use. The definition of symptoms will be:

  1. Any symptom related with intracranial hypertension, providing the patient has an Eastern cooperative Oncology Group performance status (ECOG PS) 0-2 and the other inclusion and exclusion criteria are met.
  2. Any symptom related to focal neurologic deficit.
  3. Epilepsy Note: Patients could have or not these symptoms controlled with corticosteroids at the inclusion of the clinical trial.
* A documented mutation in BRAF-V600 in the tumor tissue.
* Modified Barthel Index of Activities of Daily Living > 10 (see Appendix 5).
* Subjects aged ≥ 18 years.
* Performance status ECOG PS 0-2 (see Appendix 7).
* Able to swallowing
* Adequate hematologic function:

  1. Haemoglobin ≥ 9 g/dL (may have been transfused).
  2. Platelet count ≥ 75 × 109/L.
  3. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
* Adequate hepatic function defined by a total bilirubin level ≤ 2.0 × the upper limit of normality (ULN) and AST and ALT levels ≤ 2.5 × ULN; or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
* Serum Creatinine ≤ 2.0 x ULN or estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Immunotherapy allowed if administered in the adjuvant/neoadjuvant setting, any grade 3-4 prior toxicity must be resolved to grade 0 or at baseline levels.

Steroids or anticonvulsants are allowed if clinically needed. No dose limit of steroids is pre-specified as long as they are not in an increasing dose for the last 5 days prior to start of study treatment.

- Female subjects of childbearing potential (WOCBP) must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; refer to Appendix 8) for the duration of the study treatment and for 6 months after the last dose of study treatment.

A woman is considered of childbearing potential ( i.e. fertile) following menarche and until becoming postmenopausal unless permanently sterile. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

1. Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments
2. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the postmenopausal range
3. Radiation induced oophorectomy with last menses >1 year ago
4. Chemotherapy induced menopause with >1 year interval since last menses
5. Surgical sterilization (bilateral oophorectomy or hysterectomy)
6. Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
7. Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

   * Male study participants with WOCBP partners are required to use condoms during the study and until 6 months after the last dose of study treatment unless they are vasectomized or practice sexual abstinence.
   * WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial and until 6 months after last treatment. All men must agree not to donate sperm during the trial and for 6 months after receiving the last therapy dose.
   * Willingness and ability to attend scheduled visits, follow the treatment schedule and undergo clinical tests and other study procedures.

Exclusion Criteria:

Patients meeting any of the following criteria are excluded from the study:

* Uveal melanoma.
* History of leptomeningeal metastases unless they are a finding in the Brain MRI that does not explain the main neurological symptoms of the patient, according to physician criteria.
* Another non-cured cancer in the last 2 years, except for in situ carcinoma of the cervix, breast, prostate or squamous cell carcinoma of the skin adequately treated or limited basal cell skin cancer adequately controlled. Patients with cured cancer should be free of any adjuvant treatment (i.e chemotherapy or targeted therapy/monoclonal antibodies) with the exception of hormonal therapy for completed cured localized breast cancer or localized prostate cancer.
* History of allogeneic organ transplant.
* History of or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or history of retinal degenerative disease (RDD).
* History of interstitial lung disease.
* Systemic immunotherapy treatment for melanoma would be allowed only in the adjuvant/neoadjuvant setting (regardless if the brain relapse was during or after that) providing that ALL the following criteria are met:

  1. The immunotherapy regimen did not contain anti LAG-3 treatment.
  2. Patient did not have brain metastases (whether they were symptomatic or asymptomatic) prior to this adjuvant/neoadjuvant immunotherapy setting.
  3. Patient was treated with adjuvant/neoadjuvant for at least 6 months.
  4. No other treatments different than the one in adjuvant/neoadjuvant before symptomatic brain metastases were applied.
  5. Patient did not discontinue immunotherapy due to related adverse events.
* Targeted therapy against BRAF and/or MEK will not be allowed in any setting, including adjuvant.
* Chemotherapy will not be allowed in any setting.
* Patients in the need of urgent brain surgery before inclusion. However, patients are allowed to enter in the clinical trial after brain surgery, providing they meet the rest of inclusion and exclusion criteria, especially having at least one measurable lesion as per modified RECIST criteria after this surgery.
* Brain radiotherapy will not be allowed before entering the clinical trial. Patients can receive brain radiotherapy during the clinical trial, if they progress into the brain, as per institutional guidelines ONLY if (must fulfill the three):

  1. They have received at least TWO doses of cemiplimab and fianlimab AND
  2. The event of an intracranial progressive disease happens during cemiplimab and fianlimab AND
  3. They comply to receive encorafenib and binimetinib as rechallenge. Encorafenib and binimetinib should be stopped 24h before, during and 24h after radiotherapy.
* History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (eg, cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
* Active infection requiring therapy.
* Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
* Uncontrolled infection with HIV, HBV, or HCV infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection.

Notes:

1. Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
2. Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
3. Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
4. Patients with HIV or hepatitis must be reviewed by a qualified specialist (eg, infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial.

   * Impaired cardiovascular function or clinically significant (i.e., active) cardiovascular diseases such as: cerebrovascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), a LVEF < 50% evaluated as per institutional guidelines, or serious cardiac arrhythmia requiring medication or a triplicate average baseline QTc interval > 500 ms, history of myocarditis.

Note: Patients not fulfilling these cardiovascular criteria can be consulted to medical monitor and coordinating investigator for a case by case examination.

* TnT or troponin I TnI > 2x institutional ULN at baseline. Note: Patients with TnT or TnI levels between > 1 to 2x ULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are > 1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on the medical judgment in the patient's best interest.
* Uncontrolled arterial hypertension despite medical treatment.
* Moderate (Child Pugh Class B) or severe (Child Pugh Class C) hepatic impairment.
* Impairment of gastrointestinal function. Inability to swallow tablets or capsules.
* Neuromuscular disorders associated with high concentrations of creatine kinase.
* Subjects that have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 weeks (28 days) prior to the first dose of trial treatment, other than steroids required for brain metastasis symptoms control.
* History of pneumonitis within the last 5 years.
* Active inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis).
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
* Known hypersensitivity to the active substances or to any of the excipients.
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 5.0; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable.
* Have received a live vaccine within 30 days of planned start of study therapy. Note: Live or live attenuated vaccination with replicating potential. If a patient intends to receive a COVID-19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of study treatment.
* Known alcohol or drug abuse.
* Participation in any interventional drug or medical device study within 30 days prior to treatment start.
* Total lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
intracranial progression-free survival (icPFS) follow-up | Throughout the study period, at 12 months from the start of treatment
  Contrast enhanced brain MRI and/or color digital photography will be performed baseline and every 8 weeks (+/-1 week) up to 12 months and according to standard practice thereafter until disease progression, independently of the end of treatment (except for documentation of disease progression).

SECONDARY OUTCOMES:
Extracraneal PFS (ecPFS) follow-up | Throughout the study period, at 12 months from the start of treatment
  Body CT-scan and/or color digital photography will be performed baseline and every 8 weeks (+/-1 week) up to 12 months and according to standard practice thereafter until disease progression, independently of the end of treatment (except for documentation of disease progression).
Overall survival (OS) | Throughout the study period, at 6, 12 and 24 months from start of treatment
  Follow up at least every 4 weeks until end of study, patient withdrawal or death, whichever occurs first.
Barthel index follow-up | Throughout the study period, at weeks 8 and 24 after the start of study treatment.
  Barthel index will be monitored at baseline and at every other cycle (every 3 weeks during cemiplimab fianlimab and 4 weeks during encorafenib binimetinib) until progression.
  The Barthel Index for Activities of Daily Living is an ordinal scale which measures a person's ability to complete activities of daily living (ADL). The Barthel Index assesses the functional situation of the elderly person within a range of 0 to 100 pointss. A menor puntuación, más dependencia; y a mayor puntuación, más independencia. The lower the score, the greater thedependency; and the higher the score, the greater the independence:
  * 0-20 Total dependence
  * 21-60 Severe dependence
  * 61-90 Moderate dependence
  * 91-99 Mild dependence
  * 100 Independence
Adverse events (AE) | Throughout the study period, at 24 month from start treatment
  Adverse events (AE) assessment: type, frequency, grade, outcome, relation with study treatment (TRAE)
Serious adverse events (SAEs) assessment | Throughout the study period, at 24 month from start treatment
  Serious adverse events (SAEs) assessment: type, frequency, grade, outcome, relation with study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Marquez-Rodas, M.D., Ph.D., Study Director — Hospital General Universitario Gregorio Marañón
Locations (18):
- Spain (18):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Quiron Dexeus - IOR, Barcelona, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Instituto Catalán de Oncología - Hospital Duran i Reynals, Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos, Burgos
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario San Pedro de Alcántara, Cáceres, Cáceres
  - Onkologikoa (Donostia), Donostia / San Sebastian, Donostia
  - Hospital Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario Puerta del Hierro, Majadahonda, Madrid
  - Clinico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Regional Universitario de Málaga, Málaga, Málaga
  - Hospital Virgen de la Macarena (Sevilla), Seville, Sevilla
  - Hospital Clínico Universitario Valencia., Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez-Rodas I, Alvarez A, Arance A, Valduvieco I, Berciano-Guerrero MA, Delgado R, Soria A, Lopez Campos F, Sanchez P, Romero JL, Martin-Liberal J, Lucas A, Diaz-Beveridge R, Conde-Moreno AJ, Alamo de la Gala MDC, Garcia-Castano A, Prada PJ, Gonzalez Cao M, Puertas E, Vidal J, Foro P, Aguado de la Rosa C, Corona JA, Cerezuela-Fuentes P, Lopez P, Luna P, Aymar N, Puertolas T, Sanagustin P, Berrocal A. Encorafenib and binimetinib followed by radiotherapy for patients with BRAFV600-mutant melanoma and brain metastases (E-BRAIN/GEM1802 phase II study). Neuro Oncol. 2024 Nov 4;26(11):2074-2083. doi: 10.1093/neuonc/noae116. PMID 38946469
- [Background] Lau PKH, Feran B, Smith L, Lasocki A, Molania R, Smith K, Weppler A, Angel C, Kee D, Bhave P, Lee B, Young RJ, Iravani A, Yeang HA, Vergara IA, Kok D, Drummond K, Neeson PJ, Sheppard KE, Papenfuss T, Solomon BJ, Sandhu S, McArthur GA. Melanoma brain metastases that progress on BRAF-MEK inhibitors demonstrate resistance to ipilimumab-nivolumab that is associated with the Innate PD-1 Resistance Signature (IPRES). J Immunother Cancer. 2021 Oct;9(10):e002995. doi: 10.1136/jitc-2021-002995. PMID 34625515
- [Background] Tawbi HA, Schadendorf D, Lipson EJ, Ascierto PA, Matamala L, Castillo Gutierrez E, Rutkowski P, Gogas HJ, Lao CD, De Menezes JJ, Dalle S, Arance A, Grob JJ, Srivastava S, Abaskharoun M, Hamilton M, Keidel S, Simonsen KL, Sobiesk AM, Li B, Hodi FS, Long GV; RELATIVITY-047 Investigators. Relatlimab and Nivolumab versus Nivolumab in Untreated Advanced Melanoma. N Engl J Med. 2022 Jan 6;386(1):24-34. doi: 10.1056/NEJMoa2109970. PMID 34986285
- [Background] Panella TJ, Thomas SS, McKean M, et al: A phase 3 trial comparing fianlimab (anti-LAG-3) plus cemiplimab (anti-PD-1) to pembrolizumab in patients with completely resected high-risk melanoma. Journal of Clinical Oncology 41, no. 16_suppl (June 01, 2023) TPS9598-TPS9598.
- [Background] Baramidze A, Gogishvili M, Makharadze T, et al: A phase 3 trial of fianlimab (anti-LAG-3) plus cemiplimab (anti-PD-1) versus pembrolizumab in patients with previously untreated unresectable locally advanced or metastatic melanoma. Journal of Clinical Oncology 41, no. 16_suppl (June 01, 2023) TPS9602-TPS960
- [Background] Hamid O, Lewis KD, Weise A, McKean M, Papadopoulos KP, Crown J, Kim TM, Lee DH, Thomas SS, Mehnert J, Kaczmar J, Lakhani NJ, Kim KB, Middleton MR, Rabinowits G, Spira AI, Yushak M, Mehmi I, Fang F, Chen S, Mani J, Jankovic V, Wang F, Fiaschi N, Brennan L, Paccaly A, Masinde S, Salvati M, Fury MG, Kroog G, Lowy I, Gullo G. Phase I Study of Fianlimab, a Human Lymphocyte Activation Gene-3 (LAG-3) Monoclonal Antibody, in Combination With Cemiplimab in Advanced Melanoma. J Clin Oncol. 2024 Aug 20;42(24):2928-2938. doi: 10.1200/JCO.23.02172. Epub 2024 Jun 20. PMID 38900987
- [Background] Davies MA, Saiag P, Robert C, Grob JJ, Flaherty KT, Arance A, Chiarion-Sileni V, Thomas L, Lesimple T, Mortier L, Moschos SJ, Hogg D, Marquez-Rodas I, Del Vecchio M, Lebbe C, Meyer N, Zhang Y, Huang Y, Mookerjee B, Long GV. Dabrafenib plus trametinib in patients with BRAFV600-mutant melanoma brain metastases (COMBI-MB): a multicentre, multicohort, open-label, phase 2 trial. Lancet Oncol. 2017 Jul;18(7):863-873. doi: 10.1016/S1470-2045(17)30429-1. Epub 2017 Jun 4. PMID 28592387
- [Background] Long GV, Atkinson V, Lo S, et al: Five-year overall survival from the anti-PD1 brain collaboration (ABC Study): Randomized phase 2 study of nivolumab (nivo) or nivo+ipilimumab (ipi) in patients (pts) with melanoma brain metastases (mets). J Clin Oncol. 2021;39(15_suppl):9508-950
- [Background] Sperduto PW, Chao ST, Sneed PK, Luo X, Suh J, Roberge D, Bhatt A, Jensen AW, Brown PD, Shih H, Kirkpatrick J, Schwer A, Gaspar LE, Fiveash JB, Chiang V, Knisely J, Sperduto CM, Mehta M. Diagnosis-specific prognostic factors, indexes, and treatment outcomes for patients with newly diagnosed brain metastases: a multi-institutional analysis of 4,259 patients. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):655-61. doi: 10.1016/j.ijrobp.2009.08.025. Epub 2009 Nov 26. PMID 19942357
- [Background] Ramanujam S, Schadendorf D, Long GV. Systemic therapies for melanoma brain metastases: which drug for whom and when? Chin Clin Oncol. 2015 Jun;4(2):25. doi: 10.3978/j.issn.2304-3865.2015.06.06. PMID 26112811
- [Background] Chukwueke U, Batchelor T, Brastianos P. Management of Brain Metastases in Patients With Melanoma. J Oncol Pract. 2016 Jun;12(6):536-42. doi: 10.1200/JOP.2016.011882. PMID 27288470
- [Background] Tawbi HA, Forsyth PA, Hodi FS, Algazi AP, Hamid O, Lao CD, Moschos SJ, Atkins MB, Lewis K, Postow MA, Thomas RP, Glaspy J, Jang S, Khushalani NI, Pavlick AC, Ernstoff MS, Reardon DA, Kudchadkar R, Tarhini A, Chung C, Ritchings C, Durani P, Askelson M, Puzanov I, Margolin KA. Long-term outcomes of patients with active melanoma brain metastases treated with combination nivolumab plus ipilimumab (CheckMate 204): final results of an open-label, multicentre, phase 2 study. Lancet Oncol. 2021 Dec;22(12):1692-1704. doi: 10.1016/S1470-2045(21)00545-3. Epub 2021 Nov 10. PMID 34774225